CLINICAL TRIAL: NCT02805166
Title: The Multi-center,Open-label,Single Arm Phase IV Clinical Trial of Efficacy and Safety of PEG-rhG-CSF in Patients With Lung Cancer,Head and Neck Cancer,Colorectal Cancer,Ovarian Cancer and the Other Cancer Receiving Chemotherapy
Brief Title: PEG-rhG-CSF in Patients With Malignant Solid Tumors Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-PGC-IV-01/CSPC-PGC-IV-02
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Solid Tumors
Keywords: PEG-rhG-CSF
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim

ARMS (1):
- PEG-rhG-CSF (Experimental): patients received a single dose of 100 ug/kg of PEG-rhG-CSF(pegfilgrastim), on the basis of actual body weight, as a single subcutaneous injection on day 3 after chemotherapy.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF
  Other Names: pegfilgrastim

SUMMARY:
The purpose of this study is to estimate the safety and efficacy of PEG-rhG-CSF in patients with lung cancer,head and neck cancer,colorectal cancer,and ovarian cancer receiving multi-cycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 18 years
* diagnosis of lung cancer,head and neck cancer,colorectal cancer,ovarian cancer
* Karnofsky Performance Status ≥ 70
* life expectancy of at least 3 months
* Written informed consent are acquired

Exclusion Criteria:

* uncontrolled infection,Temperature is 38.0 ℃ or higher
* pregnancy
* Other situations that investigators consider as contra-indication for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The occurrence rate of adverse event during at least three consecutive cycles chemotherapy | up to 30 days after the patient study completion
The severity of adverse event during at least three consecutive cycles chemotherapy | up to 30 days after the patient study completion

SECONDARY OUTCOMES:
the non-occurrence rate of grade IV neutropenia (ANC <0.5 x 10^9/L)during at least three consecutive cycles chemotherapy | through the study completion,an average of 5 months
the duration of grade IV neutropenia(ANC <0.5 x 10^9/L) during at least three consecutive cycles chemotherapy | through the study completion,an average of 5 months